CLINICAL TRIAL: NCT04296292
Title: The Lived Experience of Participants in an African Randomised Trial
Acronym: LEOPARD
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); Infectious Diseases Institute, Uganda (Other); University of Zimbabwe (Other)
Responsible Party: Sponsor
Other Study IDs: 17957
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2020-09

CONDITIONS: HIV; Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AMBITION Trial Participants: Individuals who have been enrolled into the AMBITION trial
  Interventions: Other: In-depth interviews
- The next-of-kin of AMBITION Trial Participants: Individuals who have provided consent for an AMBITION trial participant who had an abnormal mental status at baseline
  Interventions: Other: In-depth interviews
- AMBITION Researchers: Individuals working on the AMBITION trial
  Interventions: Other: In-depth interviews

INTERVENTIONS:
Other: In-depth interviews — In-depth interviews following a narrative line of enquiry and direct observation at each of the research sites
  Other Names: Direct observation

SUMMARY:
There has been no previous qualitative study conducted in a low-income setting which has aimed to explore the experience of individuals who enrol into a clinical trial for the management of a life-threatening illness. The investigators plan to collect data from trial participants, their next-of-kin, and researchers working on a multi-site randomised controlled trial for the treatment of HIV-associated cryptococcal meningitis.

DETAILED DESCRIPTION:
Individuals recruited into clinical trials for life-threatening illnesses are particularly vulnerable and this is especially true in low-income settings. The decision to enrol may be influenced by existing inequalities, a poor healthcare infrastructure and the fear of death. Where patients are confused or unconscious the responsibility for this decision falls on the relatives. The objectives of this study are to learn from the experience of participants, relatives and researchers involved in a randomised controlled trial, AMBITION (ISRCTN 72509687), which is testing a novel treatment approach for HIV-associated cryptococcal meningitis and is recruiting participants from multiple sites across sub-Saharan Africa.

The investigators will collect data from trial participants and their relatives who provided consent on their behalf in Gaborone, Botswana; Kampala, Uganda and Harare, Zimbabwe. Interviews will follow a narrative approach and encourage the drawing of timelines. This will be supplemented by direct observation of the research process at each of the three recruiting hospitals. In addition, interviews will take place with researchers from the African and European institutions that form the partnership through which the trial is administered. Findings from the interviews will be prospectively fed back to the individual sites and Trial Management Group to improve the ongoing trial.

ELIGIBILITY:
AMBITION Trial Participants

Inclusion Criteria:

* Enrolled onto the AMBITION trial and has completed at least six weeks of follow-up
* Not currently confused
* Willing and able to consent to the study

Exclusion Criteria:

* Nil

The next-of-kin of AMBITION Trial Participants

Inclusion Criteria:

* Provided surrogate consent for an individual who was enrolled into the AMBITION trial
* Willing and able to consent to the study

Exclusion Criteria:

* Nil

AMBITION Researchers

Inclusion Criteria:

* Currently or previously employed on the AMBITION trial
* Willing and able to consent to the study

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals enrolled onto the AMBITION trial and individuals who provided consent for them at the Gaborone, Kampala and Harare sites.
  Researchers working on AMBITION at the Gaborone, Kampala, Harare trial sites and also in the UK or France.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Experience and views of individuals involved in the AMBITION trial | 18 months
  Interviews with AMBITION trial participants and their next-of-kin will be semi-structured and follow a loose interview guide that adopts a narrative approach to understand the experience of being diagnosed with HIV-associated cryptococcal meningitis, being approached and enrolling into the trial, undergoing invasive procedures, completing follow-up and then exiting the trial. Interviews will take place during and after the trial.
  Interviews with researchers will follow a thematic line of enquiry to understand how the trial can be improved for participants as well as how transnational research partnerships could be optimised for the benefit of researchers.
  Direct observations will help to contextualise the findings from the interviews by situating them within the clinical environment.

CONTACTS AND LOCATIONS:
Locations (3):
- Botswana Harvard AIDS Institute, Gaborone, Botswana
- Infectious Diseases Institute, Uganda, Kampala, Uganda
- University of Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided
Individual transcripts and field notes may be shared with other researchers upon request and agreement by investigators.

REFERENCES:
- [Derived] Lawrence DS, Tsholo K, Ssali A, Mupambireyi Z, Hoddinott G, Nyirenda D, Meya DB, Ndhlovu C, Harrison TS, Jarvis JN, Seeley J. The Lived Experience Of Participants in an African RandomiseD trial (LEOPARD): protocol for an in-depth qualitative study within a multisite randomised controlled trial for HIV-associated cryptococcal meningitis. BMJ Open. 2021 Apr 5;11(4):e039191. doi: 10.1136/bmjopen-2020-039191. PMID 33820784